CLINICAL TRIAL: NCT00724126
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of Rifaximin 550 mg TID in the Treatment of Subjects With Non-Constipation Irritable Bowel Syndrome
Brief Title: Rifaximin 3 Times/Day (TID) for Non-Constipation Irritable Bowel Syndrome (IBS)
Acronym: TARGET 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RFIB3008
Record Dates: First submitted 2008-07-26; First posted 2008-07-29 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Non-Constipation Irritable Bowel Syndrome
Keywords: Diarrhea; Rifaximin; IBS; Abdominal pain; Bloating
MeSH Terms: conditions — Diarrhea; Abdominal Pain | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects received placebo tablets 3 times daily for 2 weeks and were followed for 10 weeks after completion of the treatment period.
  Interventions: Drug: Placebo
- Rifaximin (Experimental): Subjects received rifaximin 550 mg tablets 3 times daily for 2 weeks and were followed for 10 weeks after completion of the treatment period.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin
  Arms: Rifaximin
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of a 14-day course of rifaximin given 3 times a day vs. placebo in providing adequate relief of IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed IBS diagnosis per Rome II criteria for diagnosis of IBS.
* Colonoscopy within 2 years as part of IBS diagnostic evaluation.
* Has active symptoms of non-constipation IBS at baseline as measured by average daily scores for abdominal pain/discomfort, bloating, and stool consistency.

Exclusion Criteria:

* Symptoms of constipation.
* History of other gastrointestinal diseases.
* Type 1 or 2 diabetes.
* Lactose intolerance not controlled by lactose-free diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Bortey, Study Director — Bausch Health Americas, Inc.
Locations (86):
- United States (86):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Tempe, Arizona
  - Anaheim, California
  - Carmichael, California
  - Chula Vista, California
  - Concord, California
  - Garden Grove, California
  - Laguna Hills, California
  - Lakewood, California
  - Los Angeles, California
  - Monterey, California
  - Orange, California
  - Roseville, California
  - San Carlos, California
  - San Francisco, California
  - Bristol, Connecticut
  - Hamden, Connecticut
  - Newark, Delaware
  - Boca Raton, Florida
  - Hollywood, Florida
  - Largo, Florida
  - New Port Richey, Florida
  - New Smyrna Beach, Florida
  - Port Orange, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Elkhart, Indiana
  - Kansas City, Kansas
  - Topeka, Kansas
  - Bowling Green, Kentucky
  - Metairie, Louisiana
  - Monroe, Louisiana
  - Baltimore, Maryland
  - Elkridge, Maryland
  - Wellesley, Massachusetts
  - Ann Arbor, Michigan
  - Troy, Michigan
  - Wyoming, Michigan
  - Mexico, Missouri
  - Sicklerville, New Jersey
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - Great Neck, New York
  - Mineola, New York
  - New York, New York
  - North Massapequa, New York
  - Pomona, New York
  - Stony Brook, New York
  - Boone, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - New Bern, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Downingtown, Pennsylvania
  - Newtown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sayre, Pennsylvania
  - Anderson, South Carolina
  - Columbia, South Carolina
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Franklin, Tennessee
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - El Paso, Texas
  - Houston, Texas
  - Lewisville, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Spokane, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Pimentel M, Lembo A, Chey WD, Zakko S, Ringel Y, Yu J, Mareya SM, Shaw AL, Bortey E, Forbes WP; TARGET Study Group. Rifaximin therapy for patients with irritable bowel syndrome without constipation. N Engl J Med. 2011 Jan 6;364(1):22-32. doi: 10.1056/NEJMoa1004409. PMID 21208106
- [Derived] Lacy BE, Chang L, Rao SSC, Heimanson Z, Sayuk GS. Rifaximin Treatment for Individual and Multiple Symptoms of Irritable Bowel Syndrome With Diarrhea: An Analysis Using New End Points. Clin Ther. 2023 Mar;45(3):198-209. doi: 10.1016/j.clinthera.2023.01.010. Epub 2023 Mar 14. PMID 36922331
- [Derived] Schoenfeld P, Pimentel M, Chang L, Lembo A, Chey WD, Yu J, Paterson C, Bortey E, Forbes WP. Safety and tolerability of rifaximin for the treatment of irritable bowel syndrome without constipation: a pooled analysis of randomised, double-blind, placebo-controlled trials. Aliment Pharmacol Ther. 2014 May;39(10):1161-8. doi: 10.1111/apt.12735. Epub 2014 Apr 3. PMID 24697851

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rifaximin
Started | 321 | 316
Completed | 302 | 301
Not Completed | 19 | 15
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Lost to Follow-up | 6 | 6
Not completed — Noncompliance | 2 | 1
Not completed — Subject randomized although ineligible | 1 | 1
Not completed — Subject had to leave vicinity of site | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was the intent-to-treat population, defined as subjects who received at least 1 dose of study drug. Two randomized subjects (1 in each group) did not receive study drug and were not included in the intent-to-treat population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rifaximin | Total
Number analyzed (Participants) | 320 | 315 | 635
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 282 | 285 | 567
  >=65 years | 37 | 30 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (14.6) | 45.9 (13.9) | 46.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 227 | 452
  Male | 95 | 88 | 183
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Black or African American | 14 | 21 | 35
  White | 302 | 282 | 584
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Had Adequate Relief of Global IBS Symptoms for at Least 2 of the 4 Weeks During the Primary Evaluation Period (ie, Weeks 3 Through 6).
Description: The primary outcome measure is assessed during the 4-week period (ie, Weeks 3 through 6) immediately following 2 weeks of treatment with study drug.
  Adequate relief of global IBS symptoms was defined as a response of "yes" to the following question, which was asked weekly (every 7 days): "In regard to all your symptoms of IBS, as compared to the way you felt before you started study medication, have you, in the past 7 days, had adequate relief of your IBS symptoms? [Yes/No]"
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Rifaximin
Number analyzed (Participants) | 320 | 315
percentage of responders | 32.2 | 40.6
Statistical Analysis 1: Comparison: Placebo vs Rifaximin; Test type: Superiority or Other; p = 0.03, Regression, Logistic; The p-value was obtained from a logistic regression model with fixed effects for treatment arm and analysis center

2. Secondary Outcome: Proportion of Subjects Who Had Adequate Relief of IBS-related Bloating for at Least 2 of the 4 Weeks During the Primary Evaluation Period (ie, Weeks 3 Through 6)
Description: The secondary outcome measure is assessed during the 4-week period (ie, Weeks 3 through 6) immediately following 2 weeks of treatment with study drug.
  Adequate relief of bloating was defined as a response of "yes" to the following question, which was asked weekly (every 7 days): "In regard to your symptom of bloating, as compared to the way you felt before you started study medication, have you, in the past 7 days, had adequate relief of your IBS symptom of bloating? [Yes/No]."
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Rifaximin
Number analyzed (Participants) | 320 | 315
percentage of responders | 31.9 | 41.0
Statistical Analysis 1: Comparison: Placebo vs Rifaximin; Test type: Superiority or Other; p = 0.02, Regression, Logistic; The p-value was obtained from a logistic regression model with fixed effects for treatment arm and analysis center

ADVERSE EVENTS:
Time Frame: 12 weeks. Adverse events were collected during the 2-week treatment period and during the 10-week follow-up period.
Description: Non-systematic (patient reports) and systematic methods (investigator examinations/laboratory tests) were used to collect adverse events. A subject reporting more than one adverse event for a particular MedDRA preferred term or system organ class was counted only once for that MedDRA preferred term or system organ class.
Arm/Group | Placebo | Rifaximin
Serious Adverse Events (participants affected / at risk) | 7/320 | 7/315
Other Adverse Events (participants affected / at risk) | 94/320 | 86/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=320) | Rifaximin (N=315)
Appendicitis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=320) | Rifaximin (N=315)
Abdominal pain (Gastrointestinal disorders) | 11 | 10
Constipation (Gastrointestinal disorders) | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 13
Nausea (Gastrointestinal disorders) | 11 | 5
Bronchitis (Infections and infestations) | 9 | 7
Nasopharyngitis (Infections and infestations) | 16 | 12
Sinusitis (Infections and infestations) | 4 | 10
Upper respiratory tract infection (Infections and infestations) | 30 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Headache (Nervous system disorders) | 26 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days